CLINICAL TRIAL: NCT01199718
Title: A Phase 1, Open-Label, Dose-Escalation, Safety, Pharmacokinetic, and Pharmacodynamic Study of CX-4945 Administered Orally to Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Study of CX-4945 in Patients With Relapsed or Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cylene Pharmaceuticals (Industry)
Responsible Party: Study Director, Cylene Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C4-09-001
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Plasmacytoma
MeSH Terms: conditions — Multiple Myeloma; Plasmacytoma | interventions — silmitasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CX-4945 (Experimental): CX-4945 oral formulation
  Interventions: Drug: CX-4945

INTERVENTIONS:
Drug: CX-4945 — CX-4945 capsules, administered orally,as escalating doses. Dose schedule: four times daily for 21 consecutive days every 28 days.

SUMMARY:
This Phase 1 study of oral CX-4945 is designed to test the safety, tolerability, and highest safe dose level of this CK2 inhibitor in patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
Elevated CK2 activity has been associated with malignant transformation and aggressive tumor growth. Over expression of CK2 has been documented in multiple types of cancers, including multiple myeloma, and inhibition of CK2 represents a potential therapeutic strategy to target a specific molecular defect perpetuating many cancers. CX-4945 has demonstrated potent inhibition of CK2 enzymatic activity. This study will evaluate the safety, pharmacokinetics, and pharmacodynamic effects of CX-4945 when administered to patients with multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Males or females at least 18 years of age
* Confirmed relapsed or refractory multiple myeloma after at least two prior lines of therapy.
* Measureable disease.
* Karnofsky Performance Status at least 60%
* Adequate liver and renal function and hematology laboratory values
* Female patients of child-bearing potential must have a negative pregnancy test.
* Signed informed consent.

Exclusion Criteria:

* Treatment with systemic cancer therapy within 21 days before screening.
* Major surgery within 4 weeks or minor surgery within 2 weeks of the start of study drug.
* Grade 3 sensory neuropathy or motor neuropathy with pain
* Concurrent severe or uncontrolled medical disease.
* Active systemic fungal, bacterial, and/or viral infection.
* Difficulty with swallowing, or an active malabsorption syndrome.
* Gastrointestinal diseases including Crohn's disease or hemorrhagic coloproctitis.
* History of gastric or small bowel surgery.
* Pregnant or nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-06 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Safety | One year (assessed at Cycle 1).
  Adverse events classified as Dose limiting toxicities. Determination of maximum tolerated dose.

SECONDARY OUTCOMES:
Pharmacokinetic and pharmacodynamic assessments. | One year - assessed throughout all cycles of participation
  Blood levels of study drug when administered in escalating doses and modulation of biomarkers for CK2.
Assess for efficacy response | One year (assessed after each cycle)
  Response assessments including M-protein levels as detailed by the International Myeloma Working Group Uniform Response Criteria.
Establish the recommended Phase 2 dose | One year

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Cylene Pharmaceuticals
Locations (6):
- United States (6):
  - Kettering, Ohio
  - Oregon Health Science University, Portland, Oregon
  - Springfield, Oregon
  - Greenville, South Carolina
  - Norfolk, Virginia
  - Yakima, Washington